CLINICAL TRIAL: NCT02322138
Title: Gastrointestinal Tolerance of Formula Supplemented With Prebiotics
Brief Title: Gastrointestinal Tolerance of Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AL14
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental 1 Infant Formula (Experimental): Milk-based infant formula without prebiotics
  Interventions: Other: Experimental 1 Infant Formula
- Experimental 2 Infant Formula (Experimental): Milk-based infant formula with prebiotics
  Interventions: Other: Experimental 2 Infant Formula
- Human Milk-Fed Reference Group (Other): Breast fed infants
  Interventions: Other: Reference Group

INTERVENTIONS:
Other: Experimental 1 Infant Formula — Ready to feed infant formula to be fed ad-libitum
  Arms: Experimental 1 Infant Formula
Other: Experimental 2 Infant Formula — Ready to feed infant formula to be fed ad-libitum
  Arms: Experimental 2 Infant Formula
Other: Reference Group — Breast fed ad libitum
  Arms: Human Milk-Fed Reference Group

SUMMARY:
The study objective is to evaluate the gastrointestinal tolerance of infant formula supplemented with prebiotics.

ELIGIBILITY:
Inclusion Criteria:

* Infant is judged to be in good health.
* Infant is a singleton from a full term birth with a gestational age of 37-42 weeks.
* Infant's birth weight was > 2490 g (~5 lbs 8 oz.).
* Infant is between 0 and 8 days of age at enrollment.
* Parent(s) confirm their intention to feed their infant the study product (formula-fed infants) or human milk (human milk-fed infants) as the sole source of nutrition for the duration of the study.
* Parent(s) confirm their intention not to administer vitamin or mineral supplements, solid foods or juices to their infant from enrollment through the duration of the study.

Exclusion Criteria:

* Adverse maternal, fetal or infant medical history that effects tolerance, growth, and/or development.
* Infants using medications, home remedies, herbal preparations, probiotics or rehydration fluids that might affect GI tolerance.
* Mother intends to use a combination of breast and formula feeding.
* Participation in another study that has not been approved as a concomitant study by AN.

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Stool Consistency Questionnaire | Baseline to 35 Days of Age
  Questionnaire

SECONDARY OUTCOMES:
Stools per Day Questionnaire | Baseline to 35 Days of Age
  Questionnaire
Feeding Spit Up Questionnaire | Baseline to 35 Days of Age
  Questionnaire
Weight | Baseline to 35 Days of Age
  Measured
Length | Baseline to 35 Days of Age
  Measured
Head Circumference | Baseline to 35 Days of Age
  Measured

CONTACTS AND LOCATIONS:
Overall Officials: Janice Kajzer, MS, RD, LD, Study Chair — Abbott Nutrition
Locations (10):
- United States (10):
  - W.O.M.B Watching Over Mothers and Babies, Tucson, Arizona
  - Clinical Research Advantage/Colorado Springs Health Partners, Colorado Springs, Colorado
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - SCORE Physician Alliance, LLC, St. Petersburg, Florida
  - Michael W. Simon, M.D., PSC, Nicholasville, Kentucky
  - Women's Clinic of Lincoln, PC., Lincoln, Nebraska
  - White Oak Family Physicians DBA Asheboro Research Associates, Asheboro, North Carolina
  - Institute of Clinical Research, Mayfield Heights, Ohio
  - The Cleveland Pediatric Research Center, LLC, Middleburg Heights, Ohio
  - Tanner Memorial Clinic, Layton, Utah